CLINICAL TRIAL: NCT04779970
Title: COntrolled Interruption of Nucleos(t)Ide Analogue Treatment in Chronic Hepatitis B Infections
Brief Title: COIN-B: COntrolled Interruption of Nucleos(t)Ide Analogue Treatment in Chronic Hepatitis B Infections
Acronym: COIN-B
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STOP: Caucasian patients (Experimental): Cessation of treatment
  Interventions: Other: Cessation of ongoing treatment
- STOP: non-Caucasian patients (Experimental): Cessation of treatment
  Interventions: Other: Cessation of ongoing treatment
- Control group (No Intervention): Standard of care follow-up

INTERVENTIONS:
Other: Cessation of ongoing treatment — Cessation of ongoing treatment
  Arms: STOP: Caucasian patients; STOP: non-Caucasian patients

SUMMARY:
In this study we will prospectively stop NA in both Caucasian and non-Caucasian patients matched for gender and age, to validate the observed host and viral parameters for future roll-out of this treatment strategy.

DETAILED DESCRIPTION:
An estimated 290 million people worldwide are chronically infected with the Hepatitis B Virus (HBV). One fourth of untreated patients develop progressive liver damage and are at risk of liver-related death, which can be prevented by treatment with Nucleos(t)ide Analogues (NA). These drugs efficiently suppress viral replication, but seroclearance of the virus, defined as loss of Hepatitis B surface Antigen (HBsAg), is predicted to require an average of 36 to 52 years of treatment. Cessation of NA after long-term viral suppression in patients without HBV seroclearance might reduce costs and may even increase the chance of subsequent HBsAg loss. We have recently shown in a retrospective multicentric international study, that Caucasian ethnicity and off-treatment viral control are associated with HBsAg loss after NA cessation. In this study we will prospectively stop NA in both Caucasian and non-Caucasian patients matched for gender and age, to validate the observed host and viral parameters for future roll-out of this treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B
* Under continuous NA treatment
* >= 18 years old and <= 75 years
* HBeAg negative at start of treatment
* HBV DNA undetectable >36 months or <100 IU/mL >48 months
* ALT <= 80 U/L

Exclusion Criteria:

* Fibrosis >F2
* Active coinfection with HCV, HDV or HIV
* Pregnancy or lactation
* Immunocompromised patients
* Ever HCC or family history of HCC
* Ever participated in HBV siRNA therapeutic trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Viral control | 72 weeks
  Number of participants with viral control after treatment cessation

SECONDARY OUTCOMES:
HBsAg loss | 72 weeks
  Number of participants with HBsAg loss after treatment cessation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Vanwolleghem, MD PhD, Study Chair — University Hospital, Antwerp
Locations (26):
- Belgium (26):
  - ASZ Aalst, Aalst
  - ZNA Stuivenberg, Antwerp
  - Antwerp University Hospital, Antwerp
  - GZA Antwerp, Antwerp
  - AZ Klina, Brasschaat
  - AZ Sint-Jan Brugge, Bruges
  - CHU Brugmann, Brussels
  - CHU Saint-Pierre, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - ULB Erasme Hospital, Brussels
  - UZ Brussels, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - ZOL Genk, Genk
  - AZ Maria Middelares Gent, Ghent
  - UZ Gent, Ghent
  - Jessa Ziekenhuizen, Hasselt
  - AZ Groeninge, Kortrijk
  - Groupe Jolimont, La Louvière
  - UZ Leuven, Leuven
  - CHC Liège, Liège
  - CHU Sart-Tilmann, Liège
  - Clinique Saint-Luc Bouge, Namur
  - AZ Damiaan, Ostend
  - AZ Delta, Roeselare
  - AZ Nikolaas, Sint-Niklaas
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request and after publication of the results

REFERENCES:
- [Derived] Furquim d'Almeida A, Vanderlinden A, Bourgeois S, Mulkay JP, Serste T, Struyve M, Deressa B, Sprengers D, de Vos M, Callens J, Shihao B, Reynaert H, Deltenre P, Janssens F, Negrin-Dastis S, Starkel P, Orlent H, Van Roey G, Verhelst X, Moreno C, Delwaide J, Van Steenkiste C, Verlinden W, Colle I, Plissonnier ML, Mukadi BK, Testoni B, Zoulim F, Matheeussen V, Vanwolleghem T. Clinical Trial: Hepatitis B Virus Genotype and a Combination of End-of-Treatment Biomarkers Predict Severe Flares After Nucleos(t)ide Analogue Cessation. Aliment Pharmacol Ther. 2026 Feb;63(3):352-361. doi: 10.1111/apt.70465. Epub 2025 Nov 19. PMID 41261561